CLINICAL TRIAL: NCT01718509
Title: The SPD489-344, Phase 3, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Dose-optimization Study to Evaluate the Efficacy, Safety, and Tolerability of SPD489 in Adults Aged 18-55 Years With Moderate to Severe Binge Eating Disorder
Brief Title: SPD489 in Adults Aged 18-55 Years With Moderate to Severe Binge Eating Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD489-344; 2012-003310-14 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD489 (Lisdexamfetamine dimesylate) (Experimental)
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 (Lisdexamfetamine dimesylate) — 50 or 70 mg administered orally, once-daily for up to 12 weeks
  Other Names: Vyvanse, Venvanse, LDX
  Arms: SPD489 (Lisdexamfetamine dimesylate)
Drug: Placebo — Administered once-daily, orally, for up to 12 weeks
  Arms: Placebo

SUMMARY:
The primary objective of the study is to demonstrate the efficacy of SPD489 compared with placebo in adults (18 55 years of age inclusive) with moderate to severe Binge Eating Disorder at Visit 8 (Weeks 11 and 12) as measured by the number of binge days (defined as days during which at least 1 binge episode occurs) per week as assessed by clinical interview based on subject diary

DETAILED DESCRIPTION:
Not Required

ELIGIBILITY:
Inclusion Criteria:

The subject cannot be enrolled in the study before all of the following inclusion criteria (including test results) are met:

1. Subject is between 18-55 years of age.
2. Subject meets the following Diagnostic and Statistical Manual of Mental Disorders Fourth Edition - Text Revision (DSM-IV-TR) criteria for a diagnosis of BED:
3. Subject has a BED diagnosis.
4. Subject's BED is of at least moderate severity with subjects reporting at least 3 binge eating days per week.
5. Female subjects must have a negative serum B-HCG pregnancy test and a negative urine pregnancy test and agree to comply with any applicable contraceptive requirements.

Exclusion Criteria:

Subjects are excluded from the study if any of the following exclusion criteria are met:

1. Subject has concurrent symptoms of bulimia nervosa or anorexia nervosa.
2. Subject is receiving psychotherapy (eg, supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) or weight loss support (eg, Weight Watchers) for BED.
3. Subject has used psychostimulants to facilitate fasting or dieting as a part of their BED.
4. Subject has a lifetime history of psychosis, mania, hypomania, dementia, or ADHD.
5. Subject is considered a suicide risk, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation.
6. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems.
7. Subject has a history of moderate or severe hypertension.
8. Subject is female and pregnant or nursing.
9. Subject has had bariatric surgery, lap bands, duodenal stents, or other procedures for weight loss.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2013-09-20 (Actual); Study Completion 2013-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (48):
- United States (45):
  - Radiant Research, Inc., Tucson, Arizona
  - Southern California Research, LLC, Beverly Hills, California
  - Scripps Clinical Research Services, La Jolla, California
  - Pharmacology Research Institute, Newport Beach, California
  - Excel Research, Inc., Oceanside, California
  - PCSD - Feighner Research, San Diego, California
  - Radiant Research, Inc., Denver, Colorado
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - American Medical Research, Oak Brook, Illinois
  - Deaconess Clinic Gateway Health Center, Newburgh, Indiana
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Potomac Grove Clinical Research Center, Gaithersburg, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Activmed Practices and Research, Haverhill, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - UMN Medical School, Dept of Psychiatry, Minneapolis, Minnesota
  - Scientella, LLA, St Louis, Missouri
  - Robert Lynn Horne, MD, LTD, Las Vegas, Nevada
  - Global Medical Inst LLC; Princeton Medical Institute, Princeton, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - CNS Clinica at the Brain Resource Center, New York, New York
  - Radiant Research, Inc., Akron, Ohio
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - The Craig and Frances Lindner Center of Hope, Mason, Ohio
  - Clinical Trials of America, Inc., Eugene, Oregon
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Oregon Center for Clinical Investigators (OCCI, Inc), Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - CRI Lifetree, Philadelphia, Pennsylvania
  - Omega Medical Reserach, Warwick, Rhode Island
  - Radiant Research, Inc., Greer, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Psychiatric Medical Associates, Plano, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - NeuroScience, Inc., Herndon, Virginia
  - Summit Research Network (Seattle), LLC, Seattle, Washington
- Germany (3):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Klinische Forschung Berlin Buch GmbH, Berlin
  - Klinische Forschung Schwerin GmbH, Schwerin

REFERENCES:
- [Result] McElroy SL, Hudson J, Ferreira-Cornwell MC, Radewonuk J, Whitaker T, Gasior M. Lisdexamfetamine Dimesylate for Adults with Moderate to Severe Binge Eating Disorder: Results of Two Pivotal Phase 3 Randomized Controlled Trials. Neuropsychopharmacology. 2016 Apr;41(5):1251-60. doi: 10.1038/npp.2015.275. Epub 2015 Sep 9. PMID 26346638
- [Derived] Robertson B, Wu J, Fant RV, Schnoll SH, McElroy SL. Assessment of Amphetamine Withdrawal Symptoms of Lisdexamfetamine Dimesylate Treatment for Adults With Binge-Eating Disorder. Prim Care Companion CNS Disord. 2020 Mar 26;22(2):19m02540. doi: 10.4088/PCC.19m02540. PMID 32237290
- [Derived] Kornstein SG, Bliss C, Kando J, Madhoo M. Clinical Characteristics and Treatment Response to Lisdexamfetamine Dimesylate Versus Placebo in Adults With Binge Eating Disorder: Analysis by Gender and Age. J Clin Psychiatry. 2019 Feb 26;80(2):18m12378. doi: 10.4088/JCP.18m12378. PMID 30817099
- [Derived] Sheehan DV, Gasior M, McElroy SL, Radewonuk J, Herman BK, Hudson J. Effects of Lisdexamfetamine Dimesylate on Functional Impairment Measured on the Sheehan Disability Scale in Adults With Moderate-to-severe Binge Eating Disorder: Results from Two Randomized, Placebo-controlled Trials. Innov Clin Neurosci. 2018 Jun 1;15(5-6):22-29. PMID 30013816
- [Derived] Citrome L, Kando JC, Bliss C. Relationships between clinical scales and binge eating days in adults with moderate to severe binge eating disorder in two Phase III studies. Neuropsychiatr Dis Treat. 2018 Feb 15;14:537-546. doi: 10.2147/NDT.S158395. eCollection 2018. PMID 29497297

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD489: 50 or 70 mg administered orally, once-daily for up to 12 weeks
Period: Overall Study
Arm/Group | PLACEBO | SPD489
Started | 195 | 195
Completed | 147 | 147
Not Completed | 48 | 48
Not completed — Lost to Follow-up | 18 | 15
Not completed — Withdrawal by Subject | 7 | 13
Not completed — Adverse Event | 5 | 7
Not completed — Other | 13 | 11
Not completed — Protocol Violation | 4 | 2
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set defined as all randomized subjects who took at least 1 dose of investigational product and had at least 1 post-baseline safety assessment. 11 subjects from Site 015, 12 subjects had not been treated, and 1 subject had been treated but did not have any safety follow-up assessments were excluded from the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | SPD489 | Total
Number analyzed (Participants) | 185 | 181 | 366
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (10.01) | 37.1 (10.00) | 37.9 (10.02)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 90 | 108 | 198
  >= 40 years | 95 | 73 | 168
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 159 | 312
  Male | 32 | 22 | 54
Region of Enrollment [Count of Participants; unit: Participants]
  GERMANY | 9 | 11 | 20
  UNITED STATES | 176 | 170 | 346

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Binge Days Per Week at Visit 8 Which Spans Weeks 11/12
Description: Binge days defined as days during which at least 1 binge episode occurred. As assessed by clinical interview based on subject binge diary.
Time Frame: Baseline and Visit 8 Which Spans Weeks 11/12
Population: The Full Analysis Set was defined as all randomized subjects who took at least 1 dose of investigational product and who had 1 post-baseline primary efficacy assessment (i.e., number of binge days per week calculated for at least 1 week).
Measure: Least Squares Mean (Standard Error); unit: Binge days per week
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
Binge days per week | -2.26 (0.137) | -3.92 (0.135)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis; Least Squares Mean Difference = -1.66, 95% CI 2-sided [-2.04 to -1.28]

2. Secondary Outcome: Percent of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Up to 12 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
percentage of participants | 42.9 [35.5 to 50.2] | 86.2 [81.1 to 91.3]
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Secondary Outcome: Percent of Participants With a 4-Week Cessation From Binge Eating
Description: 4-week cessation from binge eating is defined as no binge eating episodes for 28 consecutive days prior to the last study visit.
Time Frame: Up to 12 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
percentage of participants | 13.1 [8.1 to 18.0] | 36.2 [29.1 to 43.3]
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Secondary Outcome: Percent Change From Baseline in Body Weight (kg) at Week 12
Time Frame: Baseline and week 12
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
percentage change | -0.15 (0.353) | -5.57 (0.350)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis; Least Squares Mean Difference = -5.41, 95% CI 2-sided [-6.39 to -4.44]

5. Secondary Outcome: Change From Baseline in Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) Total Score at Week 12
Description: The Y-BOCS-BE measures the obsession of binge-eating thoughts and compulsiveness of binge-eating behaviors. The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms). Total scores range from 0 to 40. Reduction in total score indicates improvement.
Time Frame: Baseline and week 12
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
units on a scale | -7.42 (0.571) | -15.36 (0.563)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis; Least Squares Mean Difference = -7.94, 95% CI 2-sided [-9.51 to -6.36]

6. Secondary Outcome: Change From Baseline in Fasting Triglyceride Levels at Up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 153 | 156
mmol/L | 0.062 (0.0453) | -0.133 (0.0449)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p = 0.002, ANCOVA; Least Squares Mean Difference = -0.196, 95% CI 2-sided [-0.321 to -0.070]

7. Secondary Outcome: Change From Baseline In Fasting Total Cholesterol Levels at Up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 153 | 156
mmol/L | -0.126 (0.0460) | -0.204 (0.0456)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p = 0.234, ANCOVA; Least Squares Mean Difference = -0.077, 95% CI 2-sided [-0.205 to 0.050]

8. Secondary Outcome: Change From Baseline in Hemoglobin A1c Levels at Up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 154 | 156
Percent | -0.02 (0.017) | 0.01 (0.017)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p = 0.185, ANCOVA; Least Squares Mean Difference = 0.03, 95% CI 2-sided [-0.02 to 0.08]

9. Secondary Outcome: Binge Eating Response
Description: Response is based on the reduction in the number of binge eating episodes. Responses were categorized as follows: -1-week Cessation = 100% reduction in binge episodes during the preceding 7 days -Marked Reduction = 99% to 75% reduction during the time since the previous visit -Moderate Reduction = 74% to 50% reduction during the time since the previous visit -Negative to Minimal Reduction = <50% reduction during the time since the previous visit
Time Frame: Up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 142 | 145
percentage of participants
  1-week cessation | 23.9 | 55.9
  Marked reduction | 13.4 | 22.8
  Moderate reduction | 19.7 | 16.6
  Negative to minimal reduction | 43.0 | 4.8
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity is not adjusted for this secondary efficacy endpoint in this study

10. Secondary Outcome: Change From Baseline in the Number of Binge Episodes Per Week at Visit 8 Which Spans Weeks 11/12
Time Frame: Baseline and Visit 8 Which Spans Weeks 11/12
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: Binge episodes per week
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
Binge episodes per week | -3.31 (0.194) | -5.54 (0.193)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least Squares Mean Difference = -2.23, 95% CI 2-sided [-2.77 to -1.69]

11. Secondary Outcome: Change From Baseline in Eating Inventory Scores at Week 12
Description: There are 36 true/false items, 14 items on a 4-point Likert scale (1=eat rarely to 4=always), and 1 item on a 6-point Likert scale (1=eat whatever you want to 6=constantly limiting food intake). Cognitive Restraint score ranges from 0-21. Hunger score ranges from 0-14. Disinhibition score ranges from 0-16. Higher scores denote higher levels of restrained eating, disinhibited eating and predisposition to hunger.
Time Frame: Baseline and week 12
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
units on a scale
  Cognitive Restraint of Eating | 2.44 (0.352) | 3.71 (0.347)
  Disinhibition of Eating | -2.01 (0.305) | -5.61 (0.300)
  Perceived Hunger | -1.93 (0.318) | -6.14 (0.313)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Cognitive Restraint of Eating; Test type: Superiority or Other; p = 0.011, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least Squares Mean Difference = 1.27, 95% CI 2-sided [0.29 to 2.24]
Statistical Analysis 2: Comparison: PLACEBO vs SPD489; Disinhibition of Eating; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least Squares Mean Difference = -3.60, 95% CI 2-sided [-4.44 to -2.76]
Statistical Analysis 3: Comparison: PLACEBO vs SPD489; Perceived Hunger; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least Squares Mean Difference = -4.21, 95% CI 2-sided [-5.09 to -3.33]

12. Secondary Outcome: Change From Baseline in Binge Eating Scale (BES) Score at Week 12
Description: The BES is a self-reported questionnaire containing 16 items designed to assess behavioral, affective, and attitudinal components of the subjective experience of binge eating. Each item is assessed based on 1 of 4 responses, with 1 denoting that a subject has greater control over eating behavior and 4 denoting that a subject had less control over eating behavior. A total score (sum of the 16 items) may range from 16-64. A lower score indicates greater control over eating behavior.
Time Frame: Baseline and week 12
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 176 | 174
units on a scale | -8.24 (0.781) | -17.52 (0.771)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least Squares Mean Difference = -9.28, 95% CI 2-sided [-11.44 to -7.12]

13. Secondary Outcome: Change From Baseline in Frontal Systems Behavior (FrSBe) Total Score at Up to 12 Weeks
Description: The FrSBe is a 46-item self-rating scale designed to measure the neurobehavioral traits associated with the 3 primary regions of the prefrontal cortex. Subjects were asked to indicate the frequency with which they have engaged in certain behaviors using a rating scale from "1" (almost never) to "5" (almost always). Summary scores were calculated and converted to t-score. A decrease from baseline in FrSBe total score represents improvement.
Time Frame: Baseline and up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: t-scores
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 153 | 158
t-scores | -3.09 (0.655) | -4.05 (0.644)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p = 0.298, ANCOVA — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least Squares Mean Difference = -0.96, 95% CI 2-sided [-2.77 to 0.85]

14. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Mobility
Description: Quality of life was assessed using the EQ-5D-5L, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Time Frame: Up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 168 | 169
percentage of participants
  No problems in walking about | 86.9 | 91.7
  Slight problems in walking about | 8.9 | 7.1
  Moderate problems walking about | 3.0 | 0.6
  Severe problems walking about | 1.2 | 0.6
  Unable to walk about | 0 | 0

15. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Self-Care
Time Frame: Up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 168 | 169
percentage of participants
  No problems washing or dressing | 97.0 | 97.0
  Slight problems washing or dressing | 2.4 | 3.0
  Moderate problems washing or dressing | 0.6 | 0
  Severe problems washing or dressing | 0 | 0
  Unable to wash or dress | 0 | 0

16. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Usual Activities
Time Frame: Up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 168 | 169
percentage of participants
  No problems doing usual activities | 82.1 | 89.9
  Slight problems dosin usual activities | 14.3 | 8.3
  Moderate problems doing usual activities | 3.0 | 1.2
  Severe problems doing usual activities | 0.6 | 0.6
  Unable to do usual activities | 0 | 0

17. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Pain/Discomfort
Time Frame: Up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 168 | 169
percentage of participants
  No pain or discomfort | 75.6 | 76.3
  Slight pain or discomfort | 18.5 | 20.1
  Moderate pain or discomfort | 3.0 | 3.0
  Severe pain or discomfort | 3.0 | 0
  Extreme pain or discomfort | 0 | 0.6

18. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Anxiety/Depression
Time Frame: Up to 12 weeks
Population: Full Analysis Set. Not all subjects had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 168 | 169
percentage of participants
  Not anxious or depressed | 69.6 | 76.3
  Slightly anxious or depressed | 23.2 | 20.7
  Moderately anxious or depressed | 4.8 | 2.4
  Severely anxious or depressed | 1.2 | 0
  Extremely anxious or depressed | 1.2 | 0.6

19. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: Up to 12 weeks
Population: For this Outcome Measure the Safety Analysis Set is defined as all randomized subjects who took at least 1 dose of investigational product and who had at least 1 post-baseline safety assessment completed, and responded to the relevant questions for the C-SSRS. All subjects from Site 015 were excluded from the Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 183 | 179
participants
  Suicidal ideation | 0 | 0
  Suicidal behavior | 0 | 0

20. Secondary Outcome: Change in Amphetamine Cessation Symptom Assessment (ACSA) Total Score From Baseline to Week 12.
Description: ACSA scale has 16 symptom items rated on a scale from 0 (not at all) to 4 (extremely) with a possible total score range of 0 to 64. Higher scores indicate greater withdrawal symptom severity. Calculated as Baseline (Day 0) - Week 12 ACSA scores.
Time Frame: Baseline and Week 12
Population: Safety Analysis Set who completed ACSC at Baseline & Week 12 Visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 142 | 135
units on a scale | 7.0 (7.69) | 4.6 (5.83)

ADVERSE EVENTS:
Description: The Safety Analysis Set defined as all randomized subjects who took at least 1 dose of investigational product and had at least 1 follow-up safety assessment.
Arm/Group | PLACEBO | SPD489
Serious Adverse Events (participants affected / at risk) | 2/185 | 1/181
Other Adverse Events (participants affected / at risk) | 43/185 | 100/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=185) | SPD489 (N=181)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=185) | SPD489 (N=181)
Constipation (Gastrointestinal disorders) | 1 (1) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 11 (12)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 60 (60)
Nausea (Gastrointestinal disorders) | 8 (9) | 16 (17)
Fatigue (General disorders) | 9 (12) | 17 (21)
Feeling jittery (General disorders) | 0 (0) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 11 (11)
Headache (Nervous system disorders) | 16 (19) | 32 (37)
Insomnia (Psychiatric disorders) | 6 (6) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.